CLINICAL TRIAL: NCT06734403
Title: Management of Patients Who Had Urolithiasis After Bladder Augmentation in Childhood
Brief Title: Urinary Calculi After Bladder Augmentation in Children
Acronym: LITAPED
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Destinval Christelle, M.D., University Hospital, Clermont-Ferrand
Other Study IDs: M24DC1104; NCT05861024 (obsolete NCT alias)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Calculi, Urinary; Neurogenic Bladder Disorder; Spina Bifida; Child, Only
Keywords: Urinary Calculus; Bladder Augmentation; Child; Retrospective Study
MeSH Terms: conditions — Urinary Calculi; Urinary Bladder, Neurogenic; Spinal Dysraphism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ileocystoplasty: Urinary Calculi After Ileocystoplasty in Children
  Interventions: Other: Bladder Augmentation
- Sigmoidocystoplasty: Urinary Calculi After Sigmoidocystoplasty in Children
  Interventions: Other: Bladder Augmentation

INTERVENTIONS:
Other: Bladder Augmentation — Bladder Augmentation using bowel loop (ileal or sigmoid loop)

SUMMARY:
The goal of this observational study is to analyse the occurence of urinary calculi after bladder augmentation in children:

* location of the calculi (kidney or bladder)
* type of bladder augmentation with higher rate of urinary calculi and why
* Find risk factors of urinary calculi in bladder augmentation (age, sex, other bladder procedures..)

DETAILED DESCRIPTION:
Study the data of patients younger than 18 years old, who underwent a bladder augmentation, complicated by urinary calculi.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 18 years old, with urinary calculi, after bladder augmentation

Exclusion Criteria:

* Patients older than 18 years old, with urinary calculi, after bladder augmentation

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients younger than 18 years old, with urinary calculi, after bladder augmentation.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Rate of participants with urinary calculi | Through study completion, an average of 2 years
  Rate of participants with urinary calculi After bladder augmentation
Location of urinary calculi in the participants | Through study completion, an average of 2 years
  After bladder augmentation, urinary calculi can be seen on postoperative imaging such as abdominal ultrasound, CT scan, and MRI. The different locations of these calculi can be the kidneys, the ureters, the bladder, or the urethra. Each patient who has had urinary calculi will be reported, and the location of the calculi will be specified depending on the imaging results.

SECONDARY OUTCOMES:
Time frame between surgery and occurence of urinary calculi in the participants After bladder augmentation | Through study completion, an average of 2 years
  Time frame between surgery and occurence of urinary calculi in the participants After bladder augmentation
Management of urinary calculi after bladder augmentation in the participants | Through study completion, an average of 2 years
  3 main procedures help getting rid off urinary calculi: extracorporeal lithotripsy, endoscopic surgery or laparotomy. The patients were divided depending on the procedure that was used to remove the urinary calculi.
Risk factors of urinary calculi after bladder augmentation in the participants | Through study completion, an average of 2 years
  Age, sex, type of bladder augmentation...

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization the investigators won't share individual participant data